CLINICAL TRIAL: NCT00003754
Title: A Phase II Study of Thalidomide and Cyclophosphamide in Patients With Recurrent or Refractory Malignancies
Brief Title: Thalidomide and Cyclophosphamide in Treating Children With Recurrent or Refractory Childhood Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 98-088; CDR0000066878 (Registry Identifier: PDQ (Physician Data Query)); MSKCC-98088A(4); NCI-G99-1498
Record Dates: First submitted 1999-11-01; First posted 2004-04-09 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Cyclophosphamide; Thalidomide

INTERVENTIONS:
Drug: cyclophosphamide
Drug: thalidomide

SUMMARY:
RATIONALE: Thalidomide may kill tumor cells by stopping the growth of new blood vessels to the tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining thalidomide with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining thalidomide and cyclophosphamide in treating children who have recurrent or refractory childhood cancers.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy and toxic effects of thalidomide and cyclophosphamide in patients with recurrent or refractory pediatric malignancies.

OUTLINE: Patients receive oral thalidomide 4 times daily. Cyclophosphamide is administered IV over 1 hour once every 4 weeks, beginning on the same day as thalidomide. Treatment continues in the absence of unacceptable toxicity or disease progression. Tumor response is assessed every 3 months.

PROJECTED ACCRUAL: A total of 45-80 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven pediatric malignancy, except when there is appearance consistent with brainstem tumor on MRI, a tumor marker positive for germ cell tumor, or ophthalmologic diagnosis of intraocular retinoblastoma Failed conventional treatment or conventional therapy is not available Measurable disease by MRI, CT scan, biochemical tumor markers, cytology, or bone marrow examination

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Lansky 60-100% OR Karnofsky 60-100% Life expectancy: At least 6 weeks Hematopoietic: Absolute neutrophil count at least 750/mm3 (between 300-750/mm3, if due to bone marrow infiltration by malignancy) Platelet count at least 75,000/mm3 (between 20,000-75,000/mm3, if due to bone marrow infiltration by malignancy) Hepatic: Bilirubin less than 2.0 mg/dL ALT less than 3 times upper limit of normal (ULN) Renal: Creatinine less than 2 times ULN OR Creatinine clearance at least 70 mL/min Neurologic: No peripheral neuropathy grade 3 or 4 No seizure disorder in patients without CNS malignancies Other: Not pregnant or nursing Negative pregnancy tests during study and for 1 month after final dose of thalidomide Fertile patients must use effective contraception during and for at least 1 month after study

PRIOR CONCURRENT THERAPY: See Disease Characteristics No limit on the number of prior agents or regimens received Biologic therapy: Prior bone marrow transplantation allowed Chemotherapy: Recovered from prior chemotherapy No prior thalidomide Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: At least 4 weeks since prior major surgery (2 weeks for minor surgery, excluding central venous catheter placement procedures)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-09; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira Dunkel, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States